CLINICAL TRIAL: NCT05904028
Title: Home OCT-Guided Treatment Versus Treat and Extend for the Management of Neovascular AMD
Acronym: AO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol AO; UG1EY014231 (NIH)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: optical coherence tomography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Visual acuity and imaging technicians will be masked to the participant's treatment group assignment, as will the central Reading Centers. Investigators, coordinators, and participants will be unmasked to treatment group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treat and Extend (Experimental): Intravitreal injections of 6 mg faricimab on a Treat and Extend schedule
  Interventions: Drug: Intravitreal injections of 6 mg faricimab on a Treat and Extend schedule
- Home optical coherence tomography-Guided Treatment (Experimental): Intravitreal injections of 6 mg faricimab on a Home OCT-guided treatment schedule
  Interventions: Device: Intravitreal injections of 6 mg faricimab on a home optical coherence tomography-guided treatment schedule

INTERVENTIONS:
Drug: Intravitreal injections of 6 mg faricimab on a Treat and Extend schedule — Intravitreal injections of 6 mg faricimab on a Treat and Extend schedule
  Arms: Treat and Extend
Device: Intravitreal injections of 6 mg faricimab on a home optical coherence tomography-guided treatment schedule — Intravitreal injections of 6 mg faricimab on a Home OCT-guided treatment schedule
  Other Names: Home OCT
  Arms: Home optical coherence tomography-Guided Treatment

SUMMARY:
Home optical coherence tomography- guided treatment versus treat and extend for the management of neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
Treatment of Neovascular Age-Related Macular Degeneration (nAMD) with anti-vascular endothelial growth factor therapy is highly effective but is associated with considerable treatment burden and cost for patients and the healthcare system. One of the principal barriers to reducing burden and cost is that the optimal number of injections needed to achieve best visual acuity and disease control for any one person is unknown. At present, there are several algorithms that modestly reduce treatment burden, but at the expense of overtreatment in some patients and less optimal disease control in others. The lack of precision in disease management may be due in part to the low frequency of disease monitoring, which typically occurs every one to two months by standard optical coherence tomography (OCT) imaging during an office visit. Home OCT imaging allows daily disease activity monitoring and the possibility of a tailored and more personalized approach to managing neovascular AMD. To understand the role of Home OCT in clinical practice, it is essential to perform a randomized clinical trial that compares visual acuity outcomes, and visit and injection frequencies, obtained using a Home OCT-guided treatment strategy versus outcomes obtained using "Treat and Extend," the treatment algorithm widely perceived to be the most common regimen in clinical practice today.

The main objective of this study is to determine if Home OCT-guided treatment results in 1) better visual acuity outcomes and/or 2) fewer number of injections over 104 weeks compared with treat and extend (T&E) dosing for nAMD.

Procedures at the baseline visit include eligibility assessment, vision testing, ocular examination, various imaging, and test session on the in-office Home OCT device. Eligible study eyes will enter the run-in phase and receive a baseline intravitreal faricimab injection. If the non-study eye also has nAMD and needs an injection, study faricimab must be used unless the protocol chair has approved of an alternative anti-VEGF. The Notal Vision Monitoring Center must confirm adequate scan quality from the study eye prior to randomization. The Reading Center must also confirm nAMD status based on a preliminary review of baseline images. One Notal Vision confirms the screening Home OCT scans are of good quality and the Reading Center confirms nAMD criteria Is met, the participant can be randomized.

Randomization of eligible study eyes must occur within 14 days of the baseline visit. Prior to randomization, the site must call the participant to confirm they are still willing to participate and agree to follow the daily Home OCT scan requirement if randomized to the Home OCT group. Sites will also confirm the participant's understanding of the trial, willingness to accept the assigned treatment group, and commitment to the follow-up schedule, and compliance with device use.

Eyes receiving an initial faricimab injection that are not eligible for the randomization phase will have a final closeout safety visit 1 month after injection.

Eyes eligible for the randomization phase will be randomly assigned 1:1 into one of two groups to guide follow-up treatment: (1) Treat and Extend or (2) Home OCT-guided treatment. Follow-up for treatment group comparisons of vision and imaging outcomes will occur at 52- and 104-week visits. Additional visits will occur every 4-18 weeks in the T&E group. Participants assigned to the Home OCT group will self-scan daily using the Home OCT device and will only return for a visit if fluid passing the threshold for an office visit is seen on Home OCT. Follow-up visit procedures include vision testing, ocular exam, and various imaging. The primary outcomes are a comparison of mean change in visual acuity and number of injections from baseline to 104 weeks between the Home OCT vs. T&E groups (study eye only)

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 50 years
* Have the capacity to consent on his/her own behalf
* Able to successfully and independently complete at least one self-scanning session on the Home OCT device located at the enrolling clinical site
* Willing to perform once daily Home OCT monitoring tests for 2 years without significant interruption (such as travel of more than 14 days)
* Best corrected E-ETDRS visual acuity ≥24 ETDRS letters (approximately 20/320 or better (Snellen))
* Previously untreated, active MNV lesion (i.e., any intraretinal or subretinal fluid within the center 3 mm diameter circle on OCT) secondary to age-related macular degeneration
* ≥ 1 intermediate drusen (≥ 63 microns) in either eye OR late AMD (MNV or macular atrophy) in the contralateral eye

Key Exclusion Criteria for Study Eye:

* Previous treatment for MNV (intravitreal injection of any anti-VEGF or anti-VEGF/anti-Ang2 agent, or any other AMD therapy)
* Prior treatment with intravitreal injection of any anti-VEGF or anti-VEGF/anti-Ang2 agent or with macular laser for any indication
* Treatment with intravitreal corticosteroids within the last 6 months
* A condition that, in the opinion of the investigator, would preclude participation in the study or ability to complete daily Home OCT scans for 2 years (e.g., unstable medical status that may preclude successful completion of follow-up, dementia, Alzheimer's disease, uncontrollable tremors)
* MNV due to other causes, such as ocular histoplasmosis, central serous choroidopathy, or pathologic myopia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
E-ETDRS Change in Visual Acuity Letter Score | Baseline to 104 weeks
  Best-corrected visual acuity following protocol-defined refraction. Visual Acuity measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent of <20/800). Higher scores indicate better visual acuity, and lower scores indicate worse visual acuity.
Number of intravitreal injections of Faricimab (6.0 mg) in the study eye | Baseline to 104 weeks

CONTACTS AND LOCATIONS:
Locations (63):
- United States (61):
  - Kent W. Small, MD, AMC, Glendale, California
  - Loma Linda University, Loma Linda, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Southern California Desert Retina Consultants, Inc., Palm Desert, California
  - UC Davis Health Eye Center, Sacramento, California
  - Macula Retina Vitreous Institute, Torrance, California
  - Bay Area Retina Associates A Medical Group, Walnut Creek, California
  - Retina Consultants, Manchester, Connecticut
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida- Jacksonville, Jacksonville, Florida
  - Florida Retina Institute, James A. Staman, MD, PA- Jacksonville, Jacksonville, Florida
  - Argus Research Center, Inc, Naples, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Northwestern Memorial Group, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - UIC - Dept of Ophthalmology & Visual Sciences, Chicago, Illinois
  - The Trustees of Indiana University, Indianapolis, Indiana
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Clinic, P.C.- West Des Moines, West Des Moines, Iowa
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - University of Kentucky Advanced Eye Care, Lexington, Kentucky
  - Elman Retina Group, BA, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Associated Retinal Consultants, Traverse City, Michigan
  - The Retina Institute, St Louis, Missouri
  - Associated Retinal Surgeons d/b/a Mid Atlantic Retina, Cherry Hill, New Jersey
  - New York University Langone Health, New York, New York
  - Macula Care, New York, New York
  - Vitreous Retina Macula Consultants of NY - VRMNY, New York, New York
  - Retina Associates of Western NY, P.C., Rochester, New York
  - The Cleveland Clinic Foundation DBA Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Verum Research LLC, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Cascade Medical Research Institute, LLC, Springfield, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - The Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hilton Head Retina Institute, Hilton Head Island, South Carolina
  - Ophthalmology Ltd., Sioux Falls, South Dakota
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants of Texas, PA, Bellaire, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Southwest Retina Consultants, El Paso, Texas
  - Baylor College of Medicine, Baylor Eye Physicians and Surgeons, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - Retinal Consultants of Texas, San Antonio, Texas
  - The Board of Regents of the University of Wisconsin System, Madison, Wisconsin
  - Eye Clinic of Wisconsin, Wausau, Wisconsin
- Canada (2):
  - Chow Berger Koushan Medicine Professional Corporation o/a Toronto Retina Institute, North YORK, Ontario
  - University Health Network, Toronto, Ontario